CLINICAL TRIAL: NCT04960670
Title: LIMIT (LIfestyle and Microbiome InTeraction) Early Adiposity Rebound in Children
Brief Title: LIMIT Early Adiposity Rebound in Children
Acronym: LIMIT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 10062021
Record Dates: First submitted 2021-06-10; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Childhood Obesity; Life Style; Intestinal Microbiome
Keywords: childhood obesity; maternal lifestyle; gut microbiome; adiposity rebound; fetal programming; first thousand days; pregnancy; breastfeeding; children nutrition; endocrine disruptors chemicals
MeSH Terms: conditions — Pediatric Obesity; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Infant stool samples for the gut microbiota analysis
  * Maternal blood samples for nutritional status evaluation.
  * Maternal urinary samples for endocrine disruptors chemicals. All biological samples will be collected and stored at -80°C until the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyads: Mother/infant pairs will be evaluated for anthropometric parameters, prenatal (dietary/lifestyle maternal factors)/postnatal determinants (type of feeding, sleep patterns, speed of growth) before discharge and after different follow-up after birth. Infant urinary and stool samples will be collected and stored. The infant adiposity rebound will be monitored.
  Interventions: Other: Evaluation of microbiome and maternal/infant lifestyle

INTERVENTIONS:
Other: Evaluation of microbiome and maternal/infant lifestyle — Identification of the longitudinal interplay between the intestinal microbiome and infant/maternal nutritional and lifestyle habits, environmental factors exposure and anthropometric measurements, in children with adiposity rebound vs children with early adiposity rebound.

SUMMARY:
Childhood obesity is a strong predictor of adult obesity with health and economic consequences for the individual and society. Adiposity rebound (AR) is a rise in the Body Mass Index occurring between 3-7 years. Early adiposity rebound (EAR) occurs at a median age of 2 years and is a risk factor for later obesity. Events happening in "the first 1,000 days" play a role in obesity development. One of the key elements in this crucial time window is the gut microbiome, a highly dynamic organ that is sensitive to environmental exposure being linked to obesity development. Prenatal (dietary/lifestyle maternal factors and environmental exposure) and postnatal determinants (the type of feeding, sleep patterns, speed of growth) and environmental obesogenic pollutants may influence the infant microbial colonization, thus increasing the risk of EAR onset.

LIMIT will holistically identify the longitudinal interplay between the intestinal microbiome and infant/maternal nutritional and lifestyle habits, environmental factors exposure and anthropometric measurements, in children with AR vs EAR, driving new mechanistic insights to create an EAR predictive model.

The study will evaluate a group of 150 mother-infant pairs, during the first four years of life at different follow-up.

ELIGIBILITY:
* Inclusion criteria: i) Infants of both sexes born to vaginal/caesarean delivery; ii) Gestational age: 37-42 weeks; iii) Italian-speaking parent; iv) 7 Ability of the parent/guardian to give informed consent; v) Ability of the mother to answer questionnaires.
* Exclusion Criteria: i) Infants with genetic/congenital diseases; ii) Infants selected for another clinical study; iii) Infants hospitalized immediately after birth; iv) Presence of gestational diabetes; v) Presence of hyperthyroidism during pregnancy; vi) Parents refusing to sign the informed consent.

Ages: 1 Day to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother and infant pairs.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant's intestinal microbiome assessment - relative abundance | 0-48 month
  To investigate the infant's intestinal microbiome development (0-48 months) by identifying the relative abundance of the dominant microbes.
Infant's intestinal microbiome assessment - microbial diversity | 0-48 month
  To investigate the infant's intestinal microbiome development (0-48 months) by assessing the microbial diversity.
Infant's intestinal microbiome assessment - inter-individual variation | 0-48 month
  To investigate the infant's intestinal microbiome development (0-48 months) by assessing the inter-individual variation.

SECONDARY OUTCOMES:
Adiposity rebound identification | 0-48 month
  To identify adiposity rebound (AR) in children, discriminating between early AR and normal AR.
Infant intestinal microbiome and pre-gestational weight status | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and pre-gestational weight status in children showing early adiposity rebound and in those showing normal adiposity rebound. In brief, maternal height (cm) and pre-pregnancy weight will be registered to calculate pre-gestational body mass index (BMI, Kg/m2).
Infant intestinal microbiome and maternal weight gain | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and maternal weight gain (Kg) during pregnancy in children showing early adiposity rebound and in those showing normal adiposity rebound.
Infant intestinal microbiome and maternal dietary habits | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome, and maternal dietary habits in children showing early adiposity rebound and in those showing normal adiposity rebound. Dietary habits will be evaluated by using a previously validated questionnaire.
Infant intestinal microbiome and maternal physical activity | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and maternal physical activity during pregnancy in children showing early adiposity rebound and in those showing normal adiposity rebound. Physical activity will be evaluated by using a previously validated questionnaire.
Infant intestinal microbiome and mode of delivery | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and mode of delivery (vaginal delivery vs. caesarean section delivery) in children showing early adiposity rebound and in those showing normal adiposity rebound.
Infant intestinal microbiome and lactation | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and lactation (breastfeeding vs. formula feeding) in children showing early adiposity rebound and in those showing normal adiposity rebound.
Infant intestinal microbiome and maternal endocrine disruptors chemicals (EDCs) exposure | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and maternal EDCs exposure (e.g. BPA, phthalates) in children showing early adiposity rebound and in those showing normal adiposity rebound.
Infant intestinal microbiome and dietary habits | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and dietary habits in children showing early adiposity rebound and in those showing normal adiposity rebound. Infant dietary habits will be evaluated by using a previously validated questionnaire.
Infant intestinal microbiome and infant sleeping habits | 0-48 month
  To identify the longitudinal interplay between infant intestinal microbiome and sleeping habits, in children showing early adiposity rebound and in those showing normal adiposity rebound.
Predictive model | 48-60 month
  To develop a predictive model for the early adiposity rebound risk taking into consideration all maternal and infant factors previously evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Rachele De Giuseppe, PhD, Principal Investigator — University of Pavia

IPD SHARING:
Plan to Share IPD: No